CLINICAL TRIAL: NCT02674061
Title: A Phase II, Open-label, Single-arm, Multicenter Study to Evaluate Efficacy and Safety of Pembrolizumab Monotherapy in Subjects With Advanced Recurrent Ovarian Cancer (KEYNOTE-100)
Brief Title: Efficacy and Safety Study of Pembrolizumab (MK-3475) in Participants With Advanced Recurrent Ovarian Cancer (MK-3475-100/KEYNOTE-100)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-100; 2015-003338-29 (EudraCT Number); 163237 (Registry Identifier: JAPIC-CTI); MK-3475-100 (Other: Merck); KEYNOTE-100 (Other: Merck)
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Ovarian Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Pembrolizumab (Experimental): Participants in Cohort A received 0-2 prior lines of treatment for recurrent ovarian cancer (ROC; 1-3 total prior lines including front-line treatment) and will be administered pembrolizumab at a dose of 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Qualified participants who complete 35 administrations of pembrolizumab but progress after discontinuation can initiate a second course of pembrolizumab 200 mg for up to 17 cycles (up to ~1 additional year).
  Interventions: Biological: Pembrolizumab
- Cohort B: Pembrolizumab (Experimental): Participants in Cohort B received 3-5 prior lines of treatment for ROC (4-6 total prior lines including front-line treatment) and will be administered pembrolizumab at a dose of 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Qualified participants who complete 35 administrations of pembrolizumab but progress after discontinuation can initiate a second course of pembrolizumab 200 mg for up to 17 cycles (up to ~1 additional year)
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered at a dose of 200 mg via IV infusion on Day 1 of each 21-day cycle
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This study will assess the efficacy and safety of pembrolizumab (MK-3475) monotherapy in female participants with recurrent ovarian cancer (ROC) who have received up to 5 prior lines of treatment including platinum-based treatment for ROC (1 to 6 total prior lines counting front line therapy). Participants will be enrolled into two separate cohorts based on the number of prior lines of treatment received for ROC. There will be no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer
* Has received a front line platinum-based regimen (administered via either intravenous or intraperitoneal route) per local standard of care or treatment guideline following the primary or interval debulking surgery with documented disease recurrence (note: Maintenance treatment following the front line treatment is permitted and counted together as part of the front line treatment)
* Has fulfilled the following additional requirements regarding prior treatments for ROC depending on the cohort participant is to be enrolled. Each participant must have documented evidence of clinical response or disease stabilization to the last regimen received.

  * Cohort A: Has received 0 to 2 additional prior lines for treating ROC (or 1-3 total prior lines counting the front line) and must have a platinum-free interval (PFI) of ≥ 3 to 12 months if the last regimen received is a platinum-based, or a treatment-free interval (TFI) of ≥ 3 to 12 months if the last regimen received is a non-platinum-based
  * Cohort B: Has received 3 to 5 additional prior lines for treating ROC (or 4-6 total prior lines counting the front line) and must have a PFI of ≥ 3 months if the last regimen received is a platinum-based, or a TFI of ≥ 3 months if the last regimen received is a non-platinum-based
* Has measurable disease at baseline based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the central imaging vendor
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has a life expectancy of ≥16 weeks
* Has provided a tumor tissue sample either collected from prior cytoreductive surgery or fresh newly obtained tumor tissue at screening
* Has adequate organ function
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug

Exclusion Criteria:

* Is currently participating in or has participated in a clinical study and received an investigational agent or used an investigational device within 4 weeks prior to the first dose of study treatment
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the planned first dose of the study
* Has had prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to the planned first dose of the study
* Has not recovered from AEs to ≤ Grade 1 or prior treatment level due to a previously administered agent
* Has epithelial ovarian cancer (EOC) with mucinous histology subtype
* Has a known additional malignancy that progressed or required active treatment within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have stable brain metastases
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has symptoms of bowel obstruction in the past 3 months
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], tumor necrosis factor receptors OX-40 or CD137) or has participated in prior pembrolizumab (MK-3475) studies
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of the planned first dose of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Matulonis UA, Shapira-Frommer R, Santin AD, Lisyanskaya AS, Pignata S, Vergote I, Raspagliesi F, Sonke GS, Birrer M, Provencher DM, Sehouli J, Colombo N, Gonzalez-Martin A, Oaknin A, Ottevanger PB, Rudaitis V, Katchar K, Wu H, Keefe S, Ruman J, Ledermann JA. Antitumor activity and safety of pembrolizumab in patients with advanced recurrent ovarian cancer: results from the phase II KEYNOTE-100 study. Ann Oncol. 2019 Jul 1;30(7):1080-1087. doi: 10.1093/annonc/mdz135. PMID 31046082
- [Derived] Ledermann JA, Shapira-Frommer R, Santin AD, Lisyanskaya AS, Pignata S, Vergote I, Raspagliesi F, Sonke GS, Birrer M, Provencher DM, Sehouli J, Colombo N, Gonzalez-Martin A, Oaknin A, Ottevanger PB, Rudaitis V, Kobie J, Nebozhyn M, Edmondson M, Sun Y, Cristescu R, Jelinic P, Keefe SM, Matulonis UA. Molecular determinants of clinical outcomes of pembrolizumab in recurrent ovarian cancer: Exploratory analysis of KEYNOTE-100. Gynecol Oncol. 2023 Nov;178:119-129. doi: 10.1016/j.ygyno.2023.09.012. Epub 2023 Oct 18. PMID 37862791
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven participants (Cohorts A=5; B = 2) received a second course of pembrolizumab at the investigator's discretion per protocol. Response/progression or adverse events (AEs) that occurred during second course of pembrolizumab were not counted towards efficacy or safety outcome measures.
Pre-assignment Details: Per protocol, progression-free survival (PFS) by Blinded Independent Central Review, Overall Survival (OS), adverse events in all participants are from end of trial database (cutoff 18-Mar-2021). Objective Response Rate (ORR), Duration of Response (DOR), Disease Control Rate (DCR), safety outcomes, and sub-group analyses of PFS, OS are from final analysis database (cutoff 18-Sep-2019).
Groups:
- Cohort A: Pembrolizumab: Participants in Cohort A received 0-2 prior lines of treatment for recurrent ovarian cancer (ROC; 1-3 total prior lines including front-line treatment) and were administered pembrolizumab at a dose of 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Qualified participants who complete 35 administrations of pembrolizumab but progress after discontinuation can initiate a second course of pembrolizumab 200 mg for up to 17 cycles (up to ~1 additional year).
- Cohort B: Pembrolizumab: Participants in Cohort B received 3-5 prior lines of treatment for ROC (4-6 total prior lines including front-line treatment) and were administered pembrolizumab at a dose of 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Qualified participants who complete 35 administrations of pembrolizumab but progress after discontinuation can initiate a second course of pembrolizumab 200 mg for up to 17 cycles (up to ~1 additional year)
Period: Overall Study
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Started | 285 | 91
Completed | 0 | 0
Not Completed | 285 | 91
Not completed — Death | 229 | 77
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 9 | 1
Not completed — Participation in Study Discontinued by Sponsor | 44 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab | Total
Number analyzed (Participants) | 285 | 91 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (11.3) | 59.5 (9.9) | 60.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 91 | 376
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 258 | 85 | 343
  Unknown or Not Reported | 21 | 3 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 3 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 253 | 85 | 338
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in All Cohort A and Cohort B Participants
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters [SOD] of target lesions) using RECIST 1.1 based on BICR. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by BICR is reported for all participants in Cohort A and Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of participants | 8.1 [5.2 to 11.9] | 9.9 [4.6 to 17.9]

2. Primary Outcome: ORR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With Programmed Cell Death Ligand -1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on BICR. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by BICR is reported here as the ORR for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by immunohistochemistry (IHC) as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of participants | 11.6 [3.9 to 25.1] | 18.2 [5.2 to 40.3]

3. Primary Outcome: ORR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on BICR. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by BICR is reported here as the ORR for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by immunohistochemistry (IHC) as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of participants | 6.9 [2.8 to 13.8] | 10.2 [3.4 to 22.2]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 based on BICR, DOR was defined as time from first documented CR or PR until progressive disease (PD) or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is a ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by Kaplan-Meier (KM) method is reported for all participants in Cohort A and Cohort B who had a confirmed CR or PR per RECIST 1.1 by BICR.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by BICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 23 | 9
Months | 8.3 [3.9 to 35.4] | 23.6 [3.3 to 32.8]

5. Secondary Outcome: DOR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 based on BICR, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD was defined as ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10 and had a confirmed CR or PR per RECIST 1.1 by BICR.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by BICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 5 | 4
Months | 11.1 [8.3 to 20.5] | NA [5.9 to NA] — NA=Median and upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse.

6. Secondary Outcome: DOR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 based on BICR, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD was defined as ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1 and had confirmed CR or PR per RECIST 1.1 by BICR.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by BICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 7 | 5
Months | 11.1 [8.2 to 35.4] | NA [5.9 to NA] — NA=Median and upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse.

7. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or Stable Disease (SD: Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or Non-CR/Non-PD (NN: does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 based on BICR. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by BICR is reported as the DCR, analyzed by test of binomial parameter, for all participants in Cohort A and Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 22.1 [17.4 to 27.4] | 22.0 [14.0 to 31.9]

8. Secondary Outcome: DCR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 based on BICR. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by BICR is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 25.6 [13.5 to 41.2] | 31.8 [13.9 to 54.9]

9. Secondary Outcome: DCR Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 based on BICR. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by BICR is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of participants | 24.8 [16.7 to 34.3] | 22.4 [11.8 to 36.6]

10. Secondary Outcome: Progression Free Survival (PFS) Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by BICR is reported for all participants in Cohort A and Cohort B.
Time Frame: Up to ~58.8 months (through database cut-off date of 18-March-2021)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Months | 2.1 [2.1 to 2.2] | 2.1 [2.1 to 2.6]

11. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by BICR is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 6
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 23.0 [18.1 to 28.1] | 27.2 [18.2 to 36.9]

12. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by BICR is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 12
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 10.5 [7.0 to 14.8] | 13.1 [6.5 to 22.2]

13. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by BICR in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by BICR is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 18
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 5.8 [3.2 to 9.5] | 13.1 [6.5 to 22.2]

14. Secondary Outcome: PFS Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Months | 2.1 [2.1 to 4.2] | 2.1 [2.0 to 8.3]

15. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 26.9 [14.4 to 41.2] | 36.8 [17.0 to 57.0]

16. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 18.2 [7.9 to 31.9] | 16.8 [3.5 to 38.7]

17. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 9.1 [2.4 to 21.3] | 16.8 [3.5 to 38.7]

18. Secondary Outcome: PFS Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Months | 2.1 [2.1 to 2.8] | 2.1 [2.1 to 3.3]

19. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 25.5 [17.2 to 34.5] | 25.6 [14.1 to 38.8]

20. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 16.4 [9.5 to 25.0] | 11.6 [3.8 to 24.4]

21. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by BICR in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by BICR is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 9.0 [3.9 to 16.7] | 11.6 [3.8 to 24.4]

22. Secondary Outcome: ORR Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by investigator is reported as the ORR for all participants in Cohort A and Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of participants | 7.0 [4.3 to 10.6] | 8.8 [3.9 to 16.6]

23. Secondary Outcome: ORR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by investigator is reported as the ORR for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of participants | 11.6 [3.9 to 25.1] | 18.2 [5.2 to 40.3]

24. Secondary Outcome: ORR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment. ORR was analyzed by test of binomial parameter. The percentage of participants who experienced CR or PR per RECIST 1.1 by investigator is reported as the ORR for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of participants | 6.9 [2.8 to 13.8] | 12.2 [4.6 to 24.8]

25. Secondary Outcome: DOR Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is a ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by KM method is reported for all participants in Cohort A and Cohort B who had a confirmed CR or PR per RECIST 1.1 by investigator.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 20 | 8
Months | 9.1 [4.0 to 35.4] | 7.5 [4.2 to 32.9]

26. Secondary Outcome: DOR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD was defined as ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10 and had a confirmed CR or PR per RECIST 1.1 by investigator.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 5 | 4
Months | 9.8 [4.0 to 22.6] | 7.3 [4.2 to 32.9]

27. Secondary Outcome: DOR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD was defined as ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. DOR analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1 and had confirmed CR or PR per RECIST 1.1 by investigator.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 7 | 6
Months | 9.8 [4.0 to 35.4] | 7.5 [4.2 to 32.9]

28. Secondary Outcome: DCR Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 by investigator assessment. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by investigator is reported as the DCR, analyzed by test of binomial parameter, for all participants in Cohort A and Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 24.9 [20.0 to 30.4] | 17.6 [10.4 to 27.0]

29. Secondary Outcome: DCR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 by investigator assessment. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by investigator is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 25.6 [13.5 to 41.2] | 27.3 [10.7 to 50.2]

30. Secondary Outcome: DCR Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: DCR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 by investigator assessment. The percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by investigator is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of participants | 24.8 [16.7 to 34.3] | 20.4 [10.2 to 34.3]

31. Secondary Outcome: PFS Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by investigator is reported for all participants in Cohort A and Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Months | 2.1 [2.1 to 2.1] | 2.1 [2.1 to 2.3]

32. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by investigator is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 6
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 24.0 [19.2 to 29.1] | 17.8 [10.7 to 26.3]

33. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by investigator is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 12
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 7.7 [4.9 to 11.3] | 6.7 [2.7 to 13.1]

34. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by Investigator in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by investigator is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 18
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 5.0 [2.8 to 8.3] | 4.4 [1.4 to 10.1]

35. Secondary Outcome: PFS Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by investigator is reported here for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
  Per protocol PFS per RECIST 1.1 by investigator was analyzed in the subgroup of Cohort A and Cohort B participants with CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Months | 2.1 [2.1 to 4.1] | 2.2 [2.0 to 4.8]

36. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 24.2 [12.5 to 38.1] | 27.3 [11.1 to 46.4]

37. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 10.8 [3.5 to 22.8] | 13.6 [3.4 to 30.9]

38. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 5.4 [1.0 to 15.8] | 9.1 [1.6 to 25.1]

39. Secondary Outcome: PFS Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. PFS per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Months | 2.1 [2.1 to 2.2] | 2.1 [2.1 to 2.2]

40. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS Rate) at Month 6 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 24.1 [16.2 to 32.9] | 20.4 [10.5 to 32.6]

41. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS Rate) at Month 12 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 11.0 [5.7 to 18.2] | 10.2 [3.7 to 20.5]

42. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by Investigator in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. The percentage of participants with PFS (PFS Rate) at Month 18 per RECIST 1.1 by investigator is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 5.6 [1.9 to 12.3] | 6.1 [1.6 to 15.2]

43. Secondary Outcome: ORR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With Platinum-Free Interval (PFI)/Treatment-Free Interval (TFI) ≥3-6 Months
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on BICR. ORR was analyzed by test of binomial parameter. Per protocol the percentage of participants who experienced CR or PR per RECIST 1.1 by BICR is reported as the ORR for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI >3-6 months subgroup analysis of ORR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of participants | 7.9 [3.8 to 14.0] |

44. Secondary Outcome: ORR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/ TFI >6-12 Months
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on BICR. ORR was analyzed by test of binomial parameter. Per protocol the percentage of participants who experienced CR or PR per RECIST 1.1 by BICR is reported as the ORR for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of ORR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 8.7 [4.2 to 15.4] |

45. Secondary Outcome: DOR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 based on BICR, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is a ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. Per protocol DOR analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months who had a CR or PR per RECIST 1.1 by BICR. Per protocol PFI/TFI ≥3-6 months subgroup analysis of DOR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by BICR. Per protocol Cohort B was excluded from PFI/TFI subgroup DOR analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 10 | 0
Months | 8.3 [4.1 to 14.5] |

46. Secondary Outcome: DOR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: For participants who demonstrated confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 based on BICR, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is a ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. Per protocol DOR analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months who had a CR or PR per RECIST 1.1 by BICR. Per protocol PFI/TFI >6-12 months subgroup analysis of DOR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by BICR. Per protocol Cohort B was excluded from PFI/TFI subgroup DOR analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 10 | 0
Months | 4.7 [3.9 to 34.6] |

47. Secondary Outcome: DCR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: DCR was defined as the percentage of participants in the analysis population who have a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 based on BICR. Per protocol the percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by BICR is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of DCR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup DCR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of participants | 18.9 [12.5 to 26.8] |

48. Secondary Outcome: DCR Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: DCR was defined as the percentage of participants in the analysis population who have a CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage to for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (does not qualify for CR or PD) for ≥24 weeks per RECIST 1.1 based on BICR. Per protocol the percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by BICR is reported as the DCR, analyzed by test of binomial parameter, for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of DCR per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup DCR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 21.7 [14.6 to 30.4] |

49. Secondary Outcome: PFS Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. Per protocol PFS per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Months | 2.1 [2.1 to 2.1] |

50. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 6 per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Month 6
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 6.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 18.2 [11.9 to 25.5] |

51. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 12 per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Month 12
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 12.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 6.4 [2.8 to 11.9] |

52. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 18 per RECIST 1.1 by BICR was not planned or conducted in Cohort B.
Time Frame: Month 18
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 18.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 1.1 [0.1 to 5.2] |

53. Secondary Outcome: PFS Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. Per protocol PFS per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Months | 2.1 [2.1 to 2.2] |

54. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 6 per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Month 6
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 6.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 23.1 [15.7 to 31.4] |

55. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 12 per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Month 12
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 12.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 12.0 [6.4 to 19.4] |

56. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by BICR in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by BICR is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 18 per RECIST 1.1 by BICR was not planned or executed in Cohort B.
Time Frame: Month 18
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup PFS rate analysis at Month 18.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 8.0 [3.5 to 14.9] |

57. Secondary Outcome: ORR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/ TFI ≥3-6 Months
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment. ORR was analyzed by test of binomial parameter. Per protocol the percentage of participants who experienced CR or PR per RECIST 1.1 by investigator is reported as the ORR for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of ORR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of participants | 8.7 [4.4 to 15.0] |

58. Secondary Outcome: ORR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/ TFI >6-12 Months
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment. ORR was analyzed by test of binomial parameter. Per protocol the percentage of participants who experienced CR or PR per RECIST 1.1 by investigator is reported as the ORR for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of ORR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: as for outcome 44
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 5.2 [1.9 to 11.0] |

59. Secondary Outcome: DOR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. Per protocol DOR analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months who had a CR or PR per RECIST 1.1 by investigator. Per protocol PFI/TFI ≥3-6 months subgroup analysis of DOR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by investigator. Per protocol Cohort B was excluded from PFI/TFI subgroup DOR analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 11 | 0
Months | 8.4 [5.0 to 17.2] |

60. Secondary Outcome: DOR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: For participants who demonstrated confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first. DOR for participants who didn't progress or die at time of analysis was censored at last tumor assessment. Per RECIST 1.1 PD is ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. Per protocol DOR analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months who had a CR or PR per RECIST 1.1 by investigator. Per protocol PFI/TFI >6-12 months subgroup analysis of DOR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug and had CR or PR per RECIST 1.1 by investigator. Per protocol Cohort B was excluded from PFI/TFI subgroup DOR analysis. DOR for all Cohort B participants was analyzed separately and not reported here.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 6 | 0
Months | 9.7 [4.0 to 34.6] |

61. Secondary Outcome: DCR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: DCR was defined as the percentage of participants in the analysis population who have CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (doesn't qualify for CR or PD) for ≥24 weeks per RECIST 1.1 by investigator assessment. Per protocol percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by investigator is reported as DCR, analyzed by test of binomial parameter, for subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of DCR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of participants | 21.3 [14.5 to 29.4] |

62. Secondary Outcome: DCR Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: DCR was defined as the percentage of participants in the analysis population who have CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD]) or NN (doesn't qualify for CR or PD) for ≥24 weeks per RECIST 1.1 by investigator assessment. Per protocol percentage of participants who experienced CR, PR, SD or NN per RECIST 1.1 by investigator is reported as DCR, analyzed by test of binomial parameter, for subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI>6-12 months subgroup analysis of DCR per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup DCR analysis. DCR for all Cohort B participants was analyzed separately and not reported here.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of participants | 23.5 [16.1 to 32.3] |

63. Secondary Outcome: PFS Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. Per protocol PFS per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: as for outcome 49
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Months | 2.1 [2.1 to 2.1] |

64. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 6 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 6
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 20.5 [13.9 to 27.9] |

65. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 12 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 12
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 6.8 [3.2 to 12.3] |

66. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of PFS rate at Month 18 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 18
Population: as for outcome 52
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 4.0 [1.4 to 8.8] |

67. Secondary Outcome: PFS Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. PFS was analyzed by KM method. Per protocol PFS per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: as for outcome 53
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Months | 2.1 [2.1 to 2.1] |

68. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 6 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 6 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 6 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 6
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 22.6 [15.5 to 30.6] |

69. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 12 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 12 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 12 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 12
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 5.6 [2.3 to 10.9] |

70. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at Month 18 Per RECIST 1.1 by Investigator in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm. The appearance of ≥1 new lesion is also PD. Per protocol the percentage of participants with PFS (PFS rate) at Month 18 per RECIST 1.1 by investigator is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of PFS rate at Month 18 per RECIST 1.1 by investigator was not planned or executed in Cohort B.
Time Frame: Month 18
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 3.7 [1.2 to 8.5] |

71. Secondary Outcome: Overall Survival (OS) in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. OS analyzed by KM method is reported for all participants in Cohort A and Cohort B.
Time Frame: Up to ~58.8 months (through database cut-off date of 18-March-2021)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Months | 18.7 [17.0 to 22.4] | 17.6 [13.3 to 24.4]

72. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 6 in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 6 is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 6
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 82.5 [77.5 to 86.4] | 79.0 [69.0 to 86.0]

73. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 12 in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 12 is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 12
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 66.0 [60.1 to 71.1] | 66.6 [55.8 to 75.3]

74. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 18 in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 18 is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 18
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 51.3 [45.4 to 57.0] | 48.5 [37.8 to 58.4]

75. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 24 in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 24 is reported for all participants in Cohort A and Cohort B.
Time Frame: Month 24
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Percentage of Participants | 40.5 [34.7 to 46.1] | 40.6 [30.4 to 50.6]

76. Secondary Outcome: OS in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from the first dose of study drug to death due to any cause. OS analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Months | 21.9 [12.9 to 26.8] | 24.0 [14.5 to NA] — Based on the statistical model used for data analysis, upper 95% CI limit was not reached by the data cut-off date.

77. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 6 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 6 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 81.0 [65.6 to 90.0] | 95.5 [71.9 to 99.3]

78. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 12 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 12 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 69.1 [52.8 to 80.7] | 86.4 [63.4 to 95.4]

79. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 18 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 18 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥10.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥10 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 43 | 22
Percentage of Participants | 54.3 [38.1 to 67.9] | 59.1 [36.1 to 76.2]

80. Secondary Outcome: OS in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from the first dose of study drug to death due to any cause. OS analyzed by KM method is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Months | 20.6 [15.2 to 23.2] | 20.7 [13.6 to 27.4]

81. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 6 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 6 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 6
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 80.0 [70.8 to 86.6] | 87.8 [74.8 to 94.3]

82. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 12 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 12 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 12
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 65.0 [54.8 to 73.5] | 75.5 [60.9 to 85.3]

83. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 18 in Subgroup of Cohort A and Cohort B Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from the first dose of study drug to death due to any cause. The percentage of participants with OS (OS rate) at Month 18 is reported for the subgroup of participants in Cohort A and Cohort B who had a PD-L1 biomarker positive expression defined by IHC as CPS ≥1.
Time Frame: Month 18
Population: Subgroup of Cohort A and Cohort B participants with CPS ≥1 who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 101 | 49
Percentage of Participants | 52.6 [42.4 to 61.9] | 53.1 [38.3 to 65.8]

84. Secondary Outcome: OS in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol OS analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of OS was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Months | 17.2 [14.0 to 20.6] |

85. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 6 in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 6 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of OS rate at Month 6 was not planned or executed in Cohort B.
Time Frame: Month 6
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 6.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 77.7 [69.4 to 84.1] |

86. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 12 in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 12 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of OS rate at Month 12 was not planned or executed in Cohort B.
Time Frame: Month 12
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 12.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 62.5 [53.4 to 70.3] |

87. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 18 in Subgroup of Cohort A Participants With PFI/TFI ≥3-6 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 18 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) ≥3-6 months. Per protocol PFI/TFI ≥3-6 months subgroup analysis of OS rate at Month 18 was not planned or executed in Cohort B.
Time Frame: Month 18
Population: Subgroup of Cohort A participants with PFI/TFI ≥3-6 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 18.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 127 | 0
Percentage of Participants | 45.2 [36.3 to 53.8] |

88. Secondary Outcome: OS in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol OS analyzed by KM method is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of OS was not planned or executed in Cohort B.
Time Frame: Up to ~43 months (through database cut-off date of 18-September-2019)
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Months | 22.1 [15.2 to 27.9] |

89. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 6 in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 6 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of OS rate at Month 6 was not planned or executed in Cohort B.
Time Frame: Month 6
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 6.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 86.1 [78.3 to 91.2] |

90. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 12 in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 12 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of OS rate at Month 12 was not planned or executed in Cohort B.
Time Frame: Month 12
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 12.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 68.7 [59.3 to 76.3] |

91. Secondary Outcome: Percentage of Participants With OS (OS Rate) at Month 18 in Subgroup of Cohort A Participants With PFI/TFI >6-12 Months
Description: OS was defined as the time from the first dose of study drug to death due to any cause. Per protocol the percentage of participants with OS (OS rate) at Month 18 is reported for the subgroup of Cohort A participants with PFI/TFI (duration from end of treatment to disease recurrence) >6-12 months. Per protocol PFI/TFI >6-12 months subgroup analysis of OS rate at Month 18 was not planned or executed in Cohort B.
Time Frame: Month 18
Population: Subgroup of Cohort A participants with PFI/TFI >6-12 months who received ≥1 dose of study drug. Per protocol Cohort B was excluded from PFI/TFI subgroup OS rate analysis at Month 18.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 115 | 0
Percentage of Participants | 54.6 [45.0 to 63.2] |

92. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. As specified by the protocol, the number of participants who experienced at least one AE is reported here for all participants in Cohort A and Cohort B.
Time Frame: Up to ~58.8 months (through database cut-off date of 18-March-2021)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Participants | 274 | 85

93. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. As specified by the protocol, the number of participants who discontinued study treatment due to an AE is reported here for all participants in Cohort A and Cohort B.
Time Frame: Up to ~58.8 months (through database cut-off date of 18-March-2021)
Population: All participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 285 | 91
Participants | 23 | 4

ADVERSE EVENTS:
Time Frame: Up to ~58.8 months (through database cut-off date of 18-March-2021)
Description: Adverse events in all participants who received ≥1 dose of study drug. Per protocol, disease progression was not considered an AE unless considered related to study drug. Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression (NP)", "Malignant NP" and "Disease progression" not related to study drug are excluded as AEs. Seven participants received a second course of pembrolizumab per protocol and were monitored for AEs and are presented separately.
Groups:
- Cohort A: Second Course Pembrolizumab: Eligible participants in Cohort A who stopped pembrolizumab with stable disease (SD) or better but progressed after stopping study treatment initiated a second course of pembrolizumab at the investigator's discretion at the same dose and schedule (200 mg Q3W) for up to 17 cycles (up to approximately 1 additional year).
- Cohort B: Second Course Pembrolizumab: Eligible participants in Cohort B who stopped pembrolizumab with SD or better but progressed after stopping study treatment initiated a second course of pembrolizumab at the investigator's discretion at the same dose and schedule (200 mg Q3W) for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab | Cohort A: Second Course Pembrolizumab | Cohort B: Second Course Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 233/285 | 77/91 | 1/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 91/285 | 26/91 | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 260/285 | 82/91 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pembrolizumab (N=285) | Cohort B: Pembrolizumab (N=91) | Cohort A: Second Course Pembrolizumab (N=5) | Cohort B: Second Course Pembrolizumab (N=2)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaldosteronism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 9 (12) | 2 (2) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (14) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Budd-Chiari syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acinetobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 1 (2) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pembrolizumab (N=285) | Cohort B: Pembrolizumab (N=91) | Cohort A: Second Course Pembrolizumab (N=5) | Cohort B: Second Course Pembrolizumab (N=2)
Anaemia (Blood and lymphatic system disorders) | 40 (58) | 13 (18) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 19 (20) | 7 (7) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 33 (33) | 11 (14) | 0 (0) | 0 (0)
Eyelid rash (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 20 (24) | 5 (5) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 76 (90) | 20 (26) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 17 (19) | 8 (9) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 31 (47) | 7 (7) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 59 (63) | 22 (25) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 56 (85) | 20 (30) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 18 (19) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 95 (123) | 24 (30) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 14 (15) | 5 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 61 (78) | 18 (24) | 0 (0) | 0 (0)
Asthenia (General disorders) | 45 (52) | 26 (29) | 0 (0) | 0 (0)
Fatigue (General disorders) | 96 (118) | 22 (27) | 1 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 22 (30) | 4 (4) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 31 (37) | 9 (11) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 16 (20) | 5 (6) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 21 (26) | 10 (13) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (19) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (21) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 19 (23) | 3 (3) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
PCO2 increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 17 (17) | 6 (6) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 76 (84) | 14 (16) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (8) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (11) | 0 (0) | 1 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (5) | 2 (6) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (33) | 14 (23) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (28) | 10 (14) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (5) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 5 (5) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (19) | 7 (8) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 21 (22) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 25 (32) | 9 (11) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 17 (19) | 3 (4) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (44) | 13 (14) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (49) | 6 (8) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15) | 3 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (35) | 12 (16) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 27 (32) | 8 (11) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (13) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02674061/Prot_SAP_001.pdf